CLINICAL TRIAL: NCT01888653
Title: Attention-Bias Modification Treatment for PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Yuval Y Neria, Professor of Medical Psychology and Director of Trauma and PTSD, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB# 6688
Record Dates: First submitted 2013-06-25; First posted 2013-06-28 (Estimated); Results first posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-02

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: PTSD; Attention Bias to threat; Attention Bias Modification Treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comparison-Training-Program (Placebo Comparator): Placebo-training program: attention control training (ACT), is identical to the ABM protocol except that during the presentation of the trials where a threat word is presented, the probe will appear with equal frequency in the position of the threat and neutral word. Thus, neither threat nor neutral words provide information regarding the position of the target probe, and there is no contingency between the position of either threat or neutral words, and the position of the probes
  Interventions: Behavioral: Attention control training (ACT)
- Attention Biased Modification (Active Comparator): Attention-bias-modification treatment (ABM) is designed to implicitly modify patients' biased threat attendance via computerized training protocols. During each session, 240 trials (80 neutral-neutral pairs, 160 threat-neutral pairs) will be presented. On trials where participants see one neutral word and one threat word, the probe will always follow the neutral word location. Thus, although there is no specific instruction to direct attention away from threat words, on 66% of all trials (and 100% of the threat-neutral trials) the position of the neutral word will indicate the position of the target probe.
  Interventions: Behavioral: Attention Bias Modification (ABM)

INTERVENTIONS:
Behavioral: Attention Bias Modification (ABM) — The training protocol consisted of 160 trials per session with 120 angry-neutral and 40 neutral-neutral trials. Each participant was trained with an alternative set of faces to the one used in the assessment task (i.e. if measured with set A then trained with set B and vice-versa). In the ABM condition, training was contin- gent on the bias measured at pre-treatment. Specifically, for those showing a bias toward the threat, the target appeared at the neutral-face location in 100% of the threat-neutral trials, while for those showing a bias away from the threat, the target appeared at the threat-face location in 100% of the threat-neutral trials.
  Other Names: ABMT
  Arms: Attention Biased Modification
Behavioral: Attention control training (ACT) — In the ACT condition, threat- face location, probe location, and probe type were fully counter- balanced with no contingency between face valence and probe location, thus resembling the assessment task.
  Other Names: ABMT Placebo
  Arms: Comparison-Training-Program

SUMMARY:
Emerging research implicates biased attention to threat in the pathophysiology of anxiety disorders. Recent findings demonstrate significant associations between attention bias and stress vulnerability. This work has motivated the development of a novel therapy, attention-bias-modification (ABM) treatment . ABM is designed to implicitly modify patients' biased threat attendance via computerized training protocols. Emerging evidence indicates that ABM is effective in modifying threat-related attention biases and in ameliorating anxiety symptoms. However, it is unclear whether ABM is efficacious for posttraumatic stress disorder (PTSD). The present pilot study is a double blind trial that seeks to examine feasibility, acceptability, safety, efficacy, and risk/benefit ratio of ABM in individuals with PTSD. In addition this pilot study seeks to identify specific genes associated with anxiety disorders and to examine whether these can predict the success of the ABM.

DETAILED DESCRIPTION:
ABM is designed to implicitly modify patients' biased threat attendance via computerized training protocols. Emerging evidence indicates that ABM is effective in modifying threat-related attention biases and in ameliorating anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 60;
* Current DSM-IV PTSD for the last 12 months or more;
* Fluent in English and willing and able to give informed written consent and participate responsibly in the protocol;
* Attention bias toward or away from threat assessed by Dot-probe attention bias task

Exclusion Criteria:

* Current DSM-IV Axis I disorder other than PTSD.
* Patients with comorbid (i.e., secondary diagnosis of) major depressive disorder (MDD) will be allowed for enrollment if their HAM-D score doesn't exceed 25;
* Prior or current diagnosis of schizophrenia, schizoaffective disorder, organic mental disorder, bipolar disorder, or antisocial, schizotypal, and schizoid personality disorders;
* Suicidal ideation or behavior that poses a significant danger to the subject. Unstable clinical condition such that participation in a controlled trial would pose a significant danger;
* Prior participation in attention bias modification treatment (ABMT);
* Current or past history of seizure disorder (except febrile seizure in childhood);
* Currently on psychotropic medication. (excluding the use of hypnotics);
* Currently participating in formal psychotherapy. This includes:

  * psychodynamic,
  * cognitive behavioral and interpersonal therapies
* Current unstable or untreated medical illness;
* Vision loss.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Neria, PhD, Principal Investigator — Columbia University and the New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric INstitute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PTSD Program, New York State Psychiatric Institute — http://columbiapsychiatry.org/ptsd

RESULTS

PARTICIPANT FLOW:
Groups:
- Attention Biased Modification: Attention-bias-modification treatment (ABM) is designed to implicitly modify patients' biased threat attendance via computerized training protocols. During each session, 240 trials (80 neutral-neutral pairs, 160 threat-neutral pairs) will be presented. On trials where participants see one neutral word and one threat word, the probe will always follow the neutral word location. Although there is no specific instruction to direct attention away from threat words, on 66% of all trials (and 100% of the threat-neutral trials) the position of the neutral word will indicate the position of the target probe.
  Attention Bias Modification (ABM): The training protocol consisted of 160 trials per session with 120 angry-neutral and 40 neutral-neutral trials. Each participant was trained with an alternative set of faces to the one used in the assessment task (i.e. if measured with set A then trained with set B and vice-versa). In the ABM condition, training was contingent on the bias measure.
Period: Overall Study
Arm/Group | Comparison-Training-Program | Attention Biased Modification
Started | 24 | 26
Completed | 24 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Comparison-Training-Program | Attention Biased Modification | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 26 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.21 (10.29) | 34.27 (10.15) | 35.68 (10.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 10 | 9 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 50
Clinician-Administered PTSD Scale (CAPS) [Mean (Standard Deviation); unit: units on a scale] — Measures severity of posttraumatic stress disorder symptoms from 0 (least severe) to 80 (most severe)
  units on a scale | 65.00 (12.08) | 62.23 (10.39) | 63.56 (11.21)
Hamilton Rating Scale for Depression (HRSD) [Mean (Standard Deviation); unit: units on a scale] — Measures severity of depression on scale from 0 (not depressed) to 52 (most severe).
  units on a scale | 13.00 (4.82) | 11.77 (5.18) | 12.36 (5.00)
PTSD Checklist Civilian Version (PCL-C) [Mean (Standard Deviation); unit: units on a scale] — Measures severity of posttraumatic stress disorder symptoms from 0 (least severe) to 80 (most severe).
  units on a scale | 62.12 (11.16) | 57.31 (9.66) | 59.62 (10.58)
Beck Depression Inventory-II (BDI-II) [Mean (Standard Deviation); unit: units on a scale] — Measures severity of depression symptoms from 0 (mildest) to 63 (most severe).
  units on a scale | 25.87 (11.34) | 24.58 (12.36) | 25.20 (11.78)

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome: Clinician Administered PTSD Scale (CAPS)
Description: Measures severity of posttraumatic stress disorder symptoms from 0 (least severe) to 80 (most severe).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comparison-Training-Program | Attention Biased Modification
Number analyzed (Participants) | 24 | 26
units on a scale | 26.44 (16.09) | 15.96 (15.75)

2. Secondary Outcome: Secondary Outcome: PTSD Check List-Civilian (PCL-C)
Description: Measures severity of posttraumatic stress disorder symptoms from 0 (least severe) to 80 (most severe).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comparison-Training-Program | Attention Biased Modification
Number analyzed (Participants) | 24 | 26
units on a scale | 20.22 (15.07) | 7.84 (10.24)

ADVERSE EVENTS:
Time Frame: Through study completion (average 1 month).
Description: The definition of adverse event and serious adverse event does not differ from the clinicaltrials.gov definition.
Arm/Group | Comparison-Training-Program | Attention Biased Modification
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26

LIMITATIONS AND CAVEATS:
While ACT is designed to train attention control in the context of attentional threat deployment, we did not directly assess attention control, and hence cannot conclusively determine that it was indeed enhanced in the ACT group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT01888653/Prot_SAP_000.pdf